CLINICAL TRIAL: NCT07393035
Title: The Effect of School-Based Environmentally Friendly Health Practices on Adolescents' Environmental Awareness, Sensitivity, and Well-Being Levels
Brief Title: School-Based Environmentally Friendly Health Practices on Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Alime Selçuk Tosun, Associate Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024/020
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Environmental Awareness and Sensitivity
Keywords: Adolescents; Environmental attitude; Psychological well-being; Environmental literacy; Recycling
MeSH Terms: conditions — Hypersensitivity; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- School-Based Environmentally Friendly Healthy Practices (Experimental): Participants in the intervention arm received a School-Based Environmentally Friendly Healthy Practices Program consisting of seven sessions. The program aimed to improve environmental awareness and sensitivity (environmental attitudes, environmental literacy, and recycling behaviors) as well as psychological well-being. In addition to the main program, participants engaged in a rhythmic exercise program for six weeks.
  Interventions: Other: School-Based Environmentally Friendly Healthy Practices Program
- Usual Care Control Group (No Intervention): Participants in the control arm did not receive the School-Based Environmentally Friendly Healthy Practices Program. They continued their routine school activities.

INTERVENTIONS:
Other: School-Based Environmentally Friendly Healthy Practices Program — Participants in the intervention arm received a School-Based Environmentally Friendly Healthy Practices Program consisting of seven sessions. The program aimed to improve environmental awareness and sensitivity (environmental attitudes, environmental literacy, and recycling behaviors) as well as psychological well-being. In addition to the main program, participants engaged in a rhythmic exercise program for six weeks.
  Arms: School-Based Environmentally Friendly Healthy Practices

SUMMARY:
This study was conducted to investigate the effect of a school-based environmentally friendly healthy practices program implemented among adolescents on the development of environmental awareness and sensitivity (environmental attitudes, environmental literacy, and recycling behaviors) and well-being levels. This research was carried out using a parallel-group randomized controlled experimental design. The study was conducted at a Secondary School. A total of 64 students participated in the study, with 32 students in the intervention group and 32 students in the control group. The School-Based Environmentally Friendly Healthy Practices Program, consisting of seven sessions, was implemented for the students. In addition to this program, a rhythmic exercise program was applied to the students for six weeks. Data were collected using a Personal Information Form. Environmental Attitude Scale, the Recycling Scale for Secondary School Students, and the Environmental Literacy Scale. Well-being levels were evaluated using the Five-Dimensional Well-Being Model for Adolescents: the EPOCH Scale.

ELIGIBILITY:
Inclusion Criteria:

- Students enrolled in the sixth grade

Exclusion Criteria:

* Students who had participated in a similar environmental or health-related program within the past year
* Students who did not attend the program for at least two consecutive weeks - Students who requested to withdraw from the study

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Environmental Attitude Scale | At baseline and one week after completion of the intervention
  The scale assesses environmental attitudes through cognitive, affective, and psychomotor dimensions. The scale consists of cognitive, affective, and psychomotor subscales. Each subscale is treated as a separate construct in line with the multidimensional conceptualization of environmental attitude. The cognitive subscale consists of 22 items, with possible scores ranging from 22 to 110. The affective subscale includes 17 items, and scores that can be obtained from this subscale range between 17 and 85. The psychomotor subscale comprises 20 items, with minimum and maximum possible scores of 20 and 100, respectively. High scores on the subscales indicate a high level of environmental attitude.

SECONDARY OUTCOMES:
Recycling Scale for Secondary School Students | At baseline and one week after completion of the intervention
  The scale evaluates the perceptions of secondary school students regarding recycling. The scale has three subscales: participation, valuing, and contribution to the economy. The scale does not have a total score. The obtainable scores for the subscales range from 5 to 25 for the participation subscale, 5 to 25 for the valuing subscale, and 5 to 20 for the contribution to the economy subscale. A high score obtained from the three subscales indicates a high level of recycling status.
Environmental Literacy Scale | At baseline and one week after completion of the intervention
  Environmental literacy was evaluated using the Environmental Literacy Scale. The minimum score that can be obtained from the scale is 20, and the maximum score is 100. A high score obtained on the scale indicates a high level of environmental literacy.
Psychological well-being score | At baseline and one week after completion of the intervention
  Psychological well-being was assessed using the Five-Dimensional Well-Being Model for Adolescents (EPOCH Scale). The scale consists of five subscales: engagement, perseverance, optimism, connectedness and happiness. The minimum score that can be obtained from the scale is 20, and the maximum score is 100. Higher scores indicate higher levels of adolescent well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Alime Selçuk Tosun, Principal Investigator — Selcuk University, Faculty of Nursing
Locations (1):
- Şerife Akkanat Secondary School, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hwong AR, Wang M, Khan H, Chagwedera DN, Grzenda A, Doty B, Benton T, Alpert J, Clarke D, Compton WM. Climate change and mental health research methods, gaps, and priorities: a scoping review. Lancet Planet Health. 2022 Mar;6(3):e281-e291. doi: 10.1016/S2542-5196(22)00012-2. PMID 35278392